CLINICAL TRIAL: NCT04416464
Title: Quality of Life and Long-term Outcomes in Patients With Pneumonia Associated With SARS-Cov2 Infection, Survivors of Intensive Care Units: a Prospective Multicenter Cohort Study
Brief Title: Quality of Life and Patient-centered Outcomes After ICU Admission for COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Centro Hospitalar do Porto (Other); Universidade do Algarve (Other); Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Sponsor
Other Study IDs: QoL_ICU_COVID
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life; Long-term Outcomes; Coronavirus Infection; Morality; Rehospitalization
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pneumonia due to SARS-CoV-2 infection: Adult hospitalized patients with pneumonia due to proven or suspected SARS-Cov-2 infection.
  Interventions: Other: COVID-19 Pneumonia

INTERVENTIONS:
Other: COVID-19 Pneumonia — Pneumonia due to proven or suspected SARS-Cov-2 infection

SUMMARY:
Patients suffering from pneumonia due to SARS-CoV-2 infection, after admission to the Intensive Care Unit (ICU), are susceptible to development of various functional sequelae, increased risk of chronic diseases, increased mortality rates and existence of relevant impacts on their quality of life in the months and years that follow the ICU admission. The present study aims to assess the determinants of health-related quality of life and patient-centered long-term outcomes among patients recovered from SARS-COV-2 pneumonia, after discharge from the ICU, its determinants and predictors, in Portugal. It is a multicenter prospective cohort study of adult patients admitted at the ICU due to proven or suspected SARS-CoV-2 infection, included 90 days after discharge from the ICU. The primary outcome is one-year health-related quality of life assessed by the EQ-5D-3L. The secondary outcomes are all-cause mortality, rehospitalizations, return to work or study, the degree of dependence and functional capacity, symptoms of anxiety, depression and post-traumatic stress, level of physical activity and cognitive, renal and respiratory functions after ICU discharge. Investigators will collect data by means of structured telephone interviews, at a 12 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older
* Admission to the intensive care unit (ICU)
* Pneumonia due to proven or suspected SARS-CoV-2 infection

Exclusion Criteria:

* Refusal to provide consent for the study by the patient or legal guardian
* ICU length of stay less than 24 hours
* Absence of telephone contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult survivors of ICU admission and pneumonia due to proven or suspected SARS-CoV-2 infection.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life. | One-year (12 months) after ICU discharge.
  The outcome will be assessed using the Portuguese version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).

SECONDARY OUTCOMES:
Length of stay at the ICU. | The outcome will be assessed 3 months after ICU discharge (at the participant enrollment).
  Length of stay at the ICU.
Incidence of all-cause mortality | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  Incidence of all-cause mortality.
Rehospitalization. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  Rehospitalization.
Percentage of long-term ventilatory support need. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  Percentage of patients requiring oxygen therapy, non-invasive ventilation, or mechanical ventilation.
Percentage of renal replacement therapy need. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  Percentage of patients requiring any kind of renal replacement therapy.
Symptoms of anxiety and depression. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  The outcome will be assessed using the Hospital Anxiety and Depression Scale (anxiety and depression scores range from 0 to 21, with higher scores indicating worse symptoms).
Score of functional independence. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  The outcome will be assessed using the Lawton & Brody Instrumental Activities of Daily Living Scale, a score of instrumental activities of daily living (the score ranges from 0 to 8, with higher scores indicating less dependence).
Score of cognitive function. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  The outcome will be assessed using the The Montreal Cognitive Assessment (MoCA). The score ranges from 0 to 30, in 8 domains, with higher scores indicating worse symptoms.
Percentage of major cardiac events. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  Percentage of major cardiac events.
Score of Chronic obstructive pulmonary disease (COPD) | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  Score of Chronic obstructive pulmonary disease (COPD) assessed using the Portuguese version of the Clinical COPD Questionnaire (CCQ). The Clinical COPD, consisting of 10 items (each scored between 0 and 6), divided into three domains (symptoms, functional, mental). The total score is calculated by summing the scores of the individual items and dividing by 10 (the number of individual items) giving a total score between 0 and 6 with higher scores representing worse scenario.
Symptoms of posttraumatic stress disorder | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  The outcome will be assessed using the Impact Event Scale-Revised (the score ranges from 0 to 88, with higher scores indicating worse symptoms).
Utility score of health-related quality of life at 3, 6, and 9 months. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  The outcome will be assessed using the Portuguese version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).
Score of self-rated health. | The outcome will be assessed at 3, 6, 9 and 12 months after ICU discharge.
  The outcome will be assessed using the visual analogue scale of the Portuguese version of the Euroqol-5D-3L questionnaire (EQ-VAS; score range from o to 100, with higher scores indicating better self-rated health).

CONTACTS AND LOCATIONS:
Overall Officials: Luís Filipe Azevedo, Prof., Principal Investigator — Universidade do Porto
Locations (3):
- Portugal (3):
  - Centro Hospitalar de Vila Nova de Gaia / Espinho - Unidade I, Vila Nova de Gaia, Porto District
  - Centro Hospitalar Universitário de São João, Porto
  - Centro Hospitalar Universitário do Porto - Hospital de Santo António, Porto

IPD SHARING:
Plan to Share IPD: Undecided
The authors encourage interested parties to contact the corresponding author with data sharing requests, including for access to additional unpublished data.